CLINICAL TRIAL: NCT05445726
Title: Clinical Validation Study for Noninvasive Cardiopulmonary Management Device
Brief Title: ECG Validation Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Analog Device, Inc. (Other)
Collaborators: Hope Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 124-332-2022
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Comparison of test device ECG to reverence device ECG.
Who Masked: Outcomes Assessor
Masking Description: Cardiologist that interpret ECG strips to not know which strip is from the reference device and which is from the test device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Healthy (Active Comparator): Generally healthy participants that are able to participate in study procedures (i.e. laying down, sitting up, shaving chest hair for ECG/Test device placement if needed).
  Interventions: Device: CPM Device
- Atrial Fibrillation Diagnosis (Active Comparator): Participants with a diagnosis of atrial fibrillation that are able to participate in study procedures (i.e. laying down, sitting up, shaving chest hair for ECG/Test device placement if needed).
  Interventions: Device: CPM Device

INTERVENTIONS:
Device: CPM Device — CPM device used in tangent with reference ECG for validation

SUMMARY:
Subjects will be recruited and begin the study as they are identified and consent to the study. Recruiting can end when 140 subjects have initiated the study. The study does allow for additional subjects to be recruited if resources allow, leading to approximately 160 subjects. At the approximate midpoint of the study, intermediate data analysis will be performed. Enrollment will continue while this occurs. Upon arrival to the clinic on the day of the study visit, prior to the application of the reference and test devices, skin inspection of the application site will be conducted. The reference ECG device will be applied, and two initial ECGs will be taken. The precordial leads from the reference device will then be removed from the patient and the CPM Device will be applied to the participant's chest as described in the IFU materials supplied with the device (the study team will also have received training on the proper placement of the device prior to the initiation of the study). This device will be worn for the remainder of the clinic visit. On the CRF, the time that the CPM Device is placed on the chest will be denoted. The reference device and the test device will then take 2 additional ECG measurements simultaneously. During ECG measurements involving CPM device, it will be helpful to maintain silence during the entire measurement duration, as it helps the device to gather heart sounds signals without interference. The ECG results will be analyzed by certified medical personnel, where they will be asked to annotate various parameters of the ECGs. The certified medical personnel will then be asked to classify the ECGs and about the strips' clinical usability.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written, informed consent
* Individuals 18 years of age and older
* Willing and able to participate in the study procedures
* If in AF cohort: subjects must have a known diagnosis of AF

Exclusion Criteria:

* Known allergy or sensitivity to ECG electrodes or any other silicone-based electrodes
* Injury or skin disturbance in the area of the test device or reference device
* Acute myocardial infarction within 90 days of screening or other cardiovascular diseases that increases subject risk or renders data uninterpretable (by discretion of the investigator)
* Stroke or TIA within 90 days of screening
* Significant tremor that prevents subject from being still
* History of abnormal life-threatening arrhythmias (by discretion of the investigator)
* Pregnant (method of assessment at study physician's discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Baseline
  Test device AFIB detection vs reference device
Specificity | Baseline
  Test device NSR detection vs reference device

SECONDARY OUTCOMES:
Clinical equivalence | Baseline
  Test device ECG strip vs reference device

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Doust, MD, Principal Investigator — Hope Research Institute
Locations (1):
- Hope Research Institute, Phoenix, Arizona, United States